CLINICAL TRIAL: NCT05424146
Title: Enhancing the Efficacy of Evidence-Based PTSD Treatment Via Microbiota-Directed Prebiotic Supplementation
Brief Title: Efficacy of Evidence-Based PTSD Treatment Via Prebiotic Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Cures Within Reach (Other)
Responsible Party: Principal Investigator, Robin Voigt, Principal Investigator, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORA 21051205
Record Dates: First submitted 2022-06-08; First posted 2022-06-21 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Non-Prebiotic Bar Group (Placebo Comparator): This group of participants will be consuming non-prebiotic bars for the duration of the trial.
  Interventions: Behavioral: Non-Prebiotic Bar +CPT
- Prebiotic Bar Group (Active Comparator): Participants will be asked to consume prebiotic bars for the duration of the trial.
  Interventions: Dietary Supplement: Prebiotic Bar +CPT

INTERVENTIONS:
Dietary Supplement: Prebiotic Bar +CPT — Participants will be instructed to consume 1 prebiotic bar once daily for 1 week CPT. Starting week 2 they will be asked to consume 1 prebiotic bar twice daily.
  Arms: Prebiotic Bar Group
Behavioral: Non-Prebiotic Bar +CPT — Participants will be instructed to consume 1 non-prebiotic bar once daily for 1 week while receiving CPT. Starting week 2 they will be asked to consume 1 non-prebiotic bar twice daily.
  Arms: Placebo Non-Prebiotic Bar Group

SUMMARY:
Posttraumatic stress disorder (PTSD) is a debilitating psychiatric disorder, which results from exposure to traumatic events. Veterans are more than twice as likely to suffer from PTSD compared to civilians. Current interventions for the treatment of PTSD are evidence-based psychotherapies, such as Cognitive Processing Therapy (CPT). Therefore, we plan to compare Cognitive Processing Therapy (CPT) with and without a novel prebiotic bar designed to beneficially modulate the microbiota to determine the utility of this combined approach to positively impact PTSD symptoms. We will conduct a 12-week randomized, double-blind, placebo-controlled, cross-sectional trial in veterans with PTSD. Participants will be randomized to receive CPT + prebiotic or CPT + placebo. They will be provided a supply of prebiotic or non prebiotic bars for 12 weeks. At three different time points, participants will complete questionnaires and complete questionnaires and produce a stool sample ( weeks 1,2, and 12). All participants will be recruited from the two-week in-person Intensive Outpatient Program (IOP) at the Rush Road Home Program, where they will be receiving CPT.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who are participating in the Rush Road Home Program 2-week Intensive Outpatient Program (IOP) and have the ability to consent.
* Ability and willingness to consume up to two prebiotic bars daily and collect stool samples.

Exclusion Criteria:

* Active suicidality or homicidality, current engagement in significant non-suicidal self harm, history of mania or psychosis, current eating disorders, and/or current substance use that would require medical observation if discontinued.
* Gastrointestinal disease: (1) prior intestinal resection, (2) history of GI disease (except for hiatal hernia, nonproton pump inhibitor requiring gastroesophageal reflux disease, or hemorrhoids), (3) known renal disease or abnormal liver function, (4) antibiotic use within the previous 12 weeks, (5) a plan to have a major change in dietary habits during the study.
* Allergy to almonds, flax seed or coconuts

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptoms scores | 12 weeks
  PTSD symptoms will be assessed using the PTSD Checklist- Identified Patient Version (PCL-5), a 20-item self-report measure of the 20 DSM-5 symptoms of PTSD. Respondents are asked to rate how bothered they have been by each of 20 items in the past month using a Likert scale ranging from 0-4, where 0= Not at All, 1= A little Bit, 2= Moderate, 3= Quite a Bit, and 4= Extremely. These scores are summed to provide a total severity score (range = 0-80). A score of 38 is considered a provisional PTSD diagnosis, the higher the scores the worse the PTSD symptoms. This questionnaire will be administered at three-time points - week 1, week 2, and week 12 to determine the time course of PTSD symptom change. Meaningful changes in symptoms will be defined as a 10-point change in the PCL-5.
Changes in microbiota community structure & function | 12 weeks
  Stool microbiota community structure will be assessed via 16S sequencing of the V4 region to characterize the intestinal microbiota communities to the genus level. Microbiota function assessed via targeted metabolomics analysis of Short Chain Fatty Acids in stool and serum (LC-MS). Stool samples are collected at three time points- week 1, week2, and week 12 to determine the time-course change.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Voigt RM, Engen PA, Villanueva M, Bambi SA, Green SJ, Naqib A, Raeisi S, Shaikh M, Hamaker BR, Cantu-Jungles TM, Pridgen SA, Held P, Keshavarzian A. Prebiotics as an adjunct therapy for posttraumatic stress disorder: a pilot randomized controlled trial. Front Neurosci. 2025 Jan 7;18:1477519. doi: 10.3389/fnins.2024.1477519. eCollection 2024. PMID 39840022

DOCUMENTS (1):
  • Informed Consent Form (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT05424146/ICF_000.pdf